CLINICAL TRIAL: NCT04597255
Title: Reproducibility and Comparison of Digital Wavefront Sensing With Conventional Shack-Hartmann Wavefront Sensing: an Explorative Study
Brief Title: Digital Wavefront Sensing
Acronym: DWS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Doreen Schmidl [dschmidl], Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-100419
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Wavefront Aberration, Corneal; Refractive Errors
Keywords: digital wavefront sensing; optical coherence tomography
MeSH Terms: conditions — Corneal Wavefront Aberration; Refractive Errors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holographic optical coherence tomography (Experimental): Healthy phakic participants
  Interventions: Device: Holographic optical coherence tomography

INTERVENTIONS:
Device: Holographic optical coherence tomography — Descriptive wavefront analysis with holographic optical coherence tomography
  Other Names: Digital wavefront sensing; Digital aberrometry

SUMMARY:
A holographic optical coherence tomography (H-OCT) setup is used to detect the wavefront by means of phase reconstruction.

DETAILED DESCRIPTION:
H-OCT will be tested in this study for its suitability for the qualitative investigation of aberrometry. We aim to achieve a digital equivalent for wavefront calculation of the widespread analog procedure commonly used with conventional wavefront-aberrometers. The results will be compared with those from a conventional analog wavefront calculation method.

In the course of this pilot study, 20 eyes of phakic and 10 eyes of pseudophakic subjects with suspected higher order aberrations will be examined using H-OCT.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Men and women aged between 18 and 85 years
3. Normal ophthalmic findings except refractive errors or suspected higher order aberrations
4. Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

1. Hyperopia > +6 Dpt. and Myopia < -6 Dpt.
2. Known ophthalmic diseases such as age related macular degeneration, diabetic retinopathy, glaucoma, retinal detachment or previous ocular trauma and surgeries except cataract extraction
3. Participation in a clinical trial in the previous 3 weeks
4. Presence of any abnormalities preventing reliable measurements as judged by the investigator
5. Pregnancy, planned pregnancy or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative description of lower order aberrations (LOA) | 14 +/- 3 days
  Zernike terms, RMS-error, Strehl ratio
Qualitative description of higher order aberrations (HOA) | 14 +/- 3 days
  Zernike terms, root mean square error
  , Strehl ratio

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Leitgeb, Prof., Principal Investigator — Meidcal University of Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar A, Drexler W, Leitgeb RA. Subaperture correlation based digital adaptive optics for full field optical coherence tomography. Opt Express. 2013 May 6;21(9):10850-66. doi: 10.1364/OE.21.010850. PMID 23669942
- [Background] Liang J, Grimm B, Goelz S, Bille JF. Objective measurement of wave aberrations of the human eye with the use of a Hartmann-Shack wave-front sensor. J Opt Soc Am A Opt Image Sci Vis. 1994 Jul;11(7):1949-57. doi: 10.1364/josaa.11.001949. PMID 8071736
- [Background] Kumar A, Wurster LM, Salas M, Ginner L, Drexler W, Leitgeb RA. In-vivo digital wavefront sensing using swept source OCT. Biomed Opt Express. 2017 Jun 21;8(7):3369-3382. doi: 10.1364/BOE.8.003369. eCollection 2017 Jul 1. PMID 28717573